CLINICAL TRIAL: NCT00541099
Title: Evaluation of Bevacizumab and Weekly Docetaxel in Elderly (≥ 75 Years) Patients With Advanced Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Bevacizumab and Docetaxel in Treating Older Patients With Stage III or Stage IV Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Shirish M. Gadgeel, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000555019; P30CA022453 (NIH); WSU-2007-053; NCT01665443 (obsolete NCT alias)
Record Dates: First submitted 2007-10-05; First posted 2007-10-08 (Estimated); Results first posted 2014-08-21 (Estimated); Last update posted 2019-03-27 (Actual); Status verified 2014-08

CONDITIONS: Lung Cancer
Keywords: stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Bevacizumab; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Avastin & Docetaxel (Experimental): Avastin 10.0 mg/kg on days 1 and 15; Dexamethasone 4 mg evening before, morning of and evening of each dose of docetaxel; Docetaxel 35 mg/m2 on day 1, 8, 15
  Interventions: Biological: bevacizumab; Drug: docetaxel

INTERVENTIONS:
Biological: bevacizumab — Avastin 10.0 mg/kg on days 1 and 15
  Other Names: Avastin
Drug: docetaxel — Dexamethasone 4 mg evening before, morning of and evening of each dose of docetaxel.Docetaxel 35 mg/m2 on day 1, 8, 15
  Other Names: TAXOTERE®

SUMMARY:
RATIONALE: Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of tumor cells by blocking blood flow to the tumor. Drugs used in chemotherapy, such as docetaxel, also work in different ways to kill tumor cells or stop them from growing. Giving bevacizumab together with docetaxel may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving bevacizumab together with docetaxel works in treating older patients with stage III or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the proportion of elderly (≥ 75 years of age) patients with stage III or IV non-small cell lung cancer surviving for at least 6 months when treated with a combination of bevacizumab and weekly docetaxel.

Secondary

* To assess the progression-free and overall survival of patients treated with this regimen.
* To determine the response rate in patients treated with this regimen.
* To assess the toxicity of this regimen in these patients.

OUTLINE: This is a multicenter study.

Patients receive bevacizumab IV over 30-90 minutes on days 1 and 15 and docetaxel IV on days 1, 8, and 15. Treatment may repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed for 4 weeks.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Inclusion criteria:

* Histologically or cytologically confirmed non-small cell lung cancer

  * Stage III or IV disease

    * Stage III disease allowed, provided the patient is not a candidate for concurrent chemotherapy and radiotherapy
  * Mixed histology allowed, provided the biopsy has less than 50% squamous cell histology
* Measurable or evaluable disease

Exclusion criteria:

* Squamous cell histology
* Evidence of cavitation in the tumor
* Tumors in close proximity to major blood vessels
* No active, untreated brain metastases

  * More than 7 days since prior treatment for brain metastases AND no evidence of hemorrhage in the lesion
  * Stable or declining dose of steroids allowed

PATIENT CHARACTERISTICS:

Inclusion criteria:

* ECOG performance status (PS) 0-2 OR Karnofsky PS 60-100%
* Life expectancy > 12 weeks
* Leukocytes ≥ 3,000/μL
* Absolute neutrophil count ≥ 1,500/μL
* Platelet count ≥ 100,000/μL
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST and ALT ≤ 2.5 times ULN (< 5 times ULN if patients has liver metastases)
* Creatinine ≤ 1.5 times normal
* Left ventricular function ≥ normal by MUGA scan or ECHO
* Urine protein:creatinine ratio ≤ 1.0 AND/OR urine protein ≤ 1+ by dipstick analysis OR protein ≤ 1 g/24-hour urine collection
* Fertile patients must use effective contraception and women should avoid breastfeeding

Exclusion criteria:

* Resting blood pressure (BP) consistently > 140/90 mm Hg

  * Patients whose BP is controlled (≤ 140 mm Hg systolic and ≤ 90 mm Hg diastolic) after adjusting, starting, or increasing the medications are eligible
* Significant hemorrhage (i.e., > 30 mL bleeding/episode ) or hemoptysis (i.e., > 5 mL fresh blood in one episode) in the previous 3 months
* Evidence of bleeding diathesis or coagulopathy
* Significant traumatic injury within the past 28 days
* Abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 6 months
* History of other active malignancies

  * If patient has other cancers such as PSA only (without clinical or radiographic evidence) prostate cancer, the patient can still be considered for this protocol if, in the clinical judgment of the treating physician, NSCLC is the most important malignancy and the other malignancy will not impact patient's overall survival
* Myocardial infarction or cerebrovascular episode within the past year
* Serious nonhealing wound or ulcer
* Significant vascular disease such as aortic aneurysm, aortic dissection, or symptomatic peripheral vascular disease
* Uncontrolled concurrent illness that would limit compliance with study requirements including, but not limited to, the following:

  * Ongoing or active infection
  * New York Heart Association class II-IV congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness/social situations
* Known hypersensitivity to any component of bevacizumab

PRIOR CONCURRENT THERAPY:

* More than 7 days since prior radiotherapy and recovered
* No concurrent full-dose warfarin or its equivalent (i.e., unfractionated and/or low molecular-weight heparin)
* More than 10 days since prior and no concurrent aspirin ≥ 325 mg/day or chronic use of nonsteroidal anti-inflammatory drugs
* More than 28 days since prior and no concurrent major surgical procedure or open biopsy
* More than 7 days since prior core biopsy or other minor procedure, excluding placement of a vascular access device
* No other concurrent investigational agents, commercial agents, or therapies
* More than 30 days since prior participation in a trial involving an investigational agent
* No prior chemotherapy

Ages: 75 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 11 (Actual)
Dates: Start 2008-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shirish M. Gadgeel, MD, Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (3):
- United States (3):
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Nevada Cancer Institute, Las Vegas, Nevada
  - Case Comprehensive Cancer Center, Cleveland, Ohio

REFERENCES:
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — http://cancer.gov/clinicaltrials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Avastin & Docetaxel
Started | 11
Completed | 8
Not Completed | 3
Not completed — Ineligible | 3

BASELINE CHARACTERISTICS:
Arm/Group | Avastin & Docetaxel
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 79.7 (4.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Survival
Time Frame: 6 months when treated with combination of Avastin and weekly docetaxel
Measure: Number (90% Confidence Interval); unit: percentage of participants surviving
Arm/Group | Avastin & Docetaxel
Number analyzed (Participants) | 8
percentage of participants surviving | 75 [40 to 95]

2. Secondary Outcome: Progression-free Survival
Description: Progression-free survival in months via the Kaplan-Meier method
Time Frame: 6 months when treated with combination of Avastin and weekly docetaxel
Population: No patient showed a response, therefore all patients had 0 for PFS
Arm/Group | Avastin & Docetaxel
Number analyzed (Participants) | 0

3. Secondary Outcome: Overall Survival
Description: Overall survival using Kaplan-Meier method.
Time Frame: 4 weeks after removal from study or until death
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Avastin & Docetaxel
Number analyzed (Participants) | 8
months | 35.7 [1.7 to 41.3]

4. Secondary Outcome: Response Rate
Time Frame: Every 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Avastin & Docetaxel
Number analyzed (Participants) | 8
Participants | 0

5. Secondary Outcome: Toxicity According to NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0
Description: Toxicity: using the highest grade of each toxicity experienced by each patient according to NCI Common Terminology Criteria for Adverse Events (CTCAE) version 3.0.
Time Frame: 1st and 2nd week of each 21 day cycle, up to six cycles.
Measure: Number; unit: Adverse event
Arm/Group | Avastin & Docetaxel
Number analyzed (Participants) | 8
Adverse event
  Serious (grade 3 or 4) | 21
  other (grade 0, 1, or 2) | 123

ADVERSE EVENTS:
Arm/Group | Avastin & Docetaxel
Serious Adverse Events (participants affected / at risk) | 3/8
Other Adverse Events (participants affected / at risk) | 6/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Avastin & Docetaxel (N=8)
Decreased ANC (Blood and lymphatic system disorders) | 1 (1)
Decreased WBC (Blood and lymphatic system disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (4)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (8)
Hypertension (Cardiac disorders) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 2 (5)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Proteinuria (Metabolism and nutrition disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Urosepsis (Renal and urinary disorders) | 1 (1)
Perineal abscess (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Avastin & Docetaxel (N=8)
Brittle Nails (Skin and subcutaneous tissue disorders) | 1 (2)
Insomina (Psychiatric disorders) | 1 (1)
UTI (Infections and infestations) | 3 (3)
Acute Colitis (Gastrointestinal disorders) | 1 (1)
Alkaline Phosphatase (Investigations) | 1 (1)
Allergic Reaction (Immune system disorders) | 1 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (5)
Anorexia (Metabolism and nutrition disorders) | 4 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bilateral Leg Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Chest Wall Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Decreased HgB (Investigations) | 2 (7)
Decreased WBC (Investigations) | 3 (6)
Dehydration (Metabolism and nutrition disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 6 (19)
Dizziness (Nervous system disorders) | 1 (1)
Dry Skin (Skin and subcutaneous tissue disorders) | 1 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (3)
epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Eye Tearing (Eye disorders) | 1 (1)
Fatigue (General disorders) | 6 (16)
Flushing (Vascular disorders) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (5)
Hemoglobin (Investigations) | 1 (5)
HTN (Vascular disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (8)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (3)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 (15)
Hyponatremia (Metabolism and nutrition disorders) | 1 (2)
Hypotension (Vascular disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Increased Creatinine (Investigations) | 1 (2)
Lacrimation (Eye disorders) | 1 (1)
Leukocytes (Blood and lymphatic system disorders) | 1 (1)
Lower Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Lymphopenia (Investigations) | 1 (6)
Metallic taste (Gastrointestinal disorders) | 1 (1)
Mucositis (Gastrointestinal disorders) | 1 (1)
Nail Changes (Skin and subcutaneous tissue disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (3)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Nose Bleed (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Oral Thrush (Gastrointestinal disorders) | 1 (1)
Pain: Chest/Torax NOS (General disorders) | 1 (2)
Pericardial Effusion (Cardiac disorders) | 1 (1)
pain: Trauma site (Injury, poisoning and procedural complications) | 1 (1)
Proteinuria (Renal and urinary disorders) | 3 (7)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (2)
R. Arm Extravasation (General disorders) | 1 (1)
R. Elbow-Soft Tissue Trauma (Injury, poisoning and procedural complications) | 1 (3)
Sensory Neuropathy (Nervous system disorders) | 2 (2)
Sinus Congest (Reproductive system and breast disorders) | 1 (1)
Sinus Drainage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Skin peeling-hands (Skin and subcutaneous tissue disorders) | 1 (1)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Taste Alteration (Gastrointestinal disorders) | 4 (6)
Tearing in eyes (Eye disorders) | 1 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
upper resp infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Urinary Frequency (Renal and urinary disorders) | 1 (2)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Vasovagal episode (Nervous system disorders) | 1 (2)
Vomiting (Gastrointestinal disorders) | 1 (3)
Watery Eye (Eye disorders) | 1 (1)
Weight Loss (Investigations) | 2 (5)
Edema: limbs (Gastrointestinal disorders) | 1 (1)
Edema: trunk/genital (Gastrointestinal disorders) | 1 (1)
Arm Laceration (General disorders) | 1 (1)
Decubitus (General disorders) | 1 (2)
Hypertension (Vascular disorders) | 3 (3)
Leukpenia (Blood and lymphatic system disorders) | 1 (2)

LIMITATIONS AND CAVEATS:
The increased use of pemetrexed in the front line setting affected accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No